CLINICAL TRIAL: NCT05212194
Title: The Relationship Between Post Dural Puncture Headache and Joint Laxity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Nezir Yılmaz, Principal investigator, Adiyaman University Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/10-25
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post spinal puncture headache (Other): the patients who developed post spinal puncture headache
  Interventions: Other: examination

INTERVENTIONS:
Other: examination — Joint laxity is scored according to the level of motion in 5 different joints and a maximum of 9 points is obtained.
  Other Names: joint laxity examination

SUMMARY:
Post-spinal headache is divided into 3 according to the severity scale. It is divided into 3 groups as mild, moderate and severe according to the presence of symptoms such as nausea, vomiting, and dizziness that prevent daily activity.

It has been reported that CSF leakage may be higher due to the weakness of the regional dural sac in primary connective tissue diseases with joint laxity and isolated joint hypermobility. Joint laxity is scored according to the level of motion in 5 different joints and a maximum of 9 points is obtained.

In this study, it was aimed to investigate whether joint laxity contributes to the development of post-spinal headache by questioning the correlation between joint laxity examination score and postspinal headache in patients with post-spinal headache.

DETAILED DESCRIPTION:
Post dural puncture headache (PDPH), also known as post lumbar puncture (LP) headache, is a common complication of diagnostic LP. It also can occur following spinal anesthesia or, more commonly, inadvertent dural puncture during attempted epidural catheter placement. The headache is usually positional (worse when upright, better when lying flat) and is often accompanied by neck stiffness, photophobia, nausea, or subjective hearing symptoms.

In various studies, common patient risk factors for PDPH have included female gender, pregnancy, age 18 to 50 years compared with older or younger ages, and a prior history of headache

Additionally it has been thought that joint laxity contributes to the development of post dural puncture headache. However, no study has been found in the literature examining this relationship between them. In thıs study it was aimed to investigate the relationship between joint laxity and post dural puncture headache.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 age
* the patients who develop PDPH

Exclusion Criteria:

* <18 and >65 age
* the patients refused to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Post dural puncture headache (PDPH) severity | 24 hours after spinal anesthesia
  The patients that occured PDPH will evaluate and classificate as mild,moderate and severe according to severity of PDPH by using Lybecker classification.
joint laxity score | 24 hours after spinal anesthesia
  The Beighton score is a simple system to quantify joint laxity and hypermobility. It uses a simple 9 point system, where the higher the score the higher the laxity.

CONTACTS AND LOCATIONS:
Overall Officials: Nezir yılmaz, Dr, Principal Investigator — Adiyaman Training and Research Hospital; Mustafa Çukurlu, Dr, Study Director — Adiyaman Training and Research Hospital
Locations (1):
- Adıyaman Training and Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No